CLINICAL TRIAL: NCT02171403
Title: Comparison of the Colonic Metabolism in Patients With Lactose Intolerance and Healthy Controls
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor Kristin Verbeke, KU Leuven
Other Study IDs: B322201421130; ML10399 (Other: UZ Leuven ethical committee)
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Lactose intolerance: Patients with a positive lactose-breath test and complaints during the test
- Lactose malabsorption: Patients with a positive lactose-breath test and no complaints during the test
- Healthy controls: Subjects with a negative lactose-breath test

SUMMARY:
Most people are born with the ability to digest lactose, a dissacharide consisting of β-D-glucose and β-D-galactose, because of the presence of lactase at the brush border of the small intestine. In about 75% of the world population the activity of this enzyme decreases after weaning (primary hypolactasia or lactase-nonpersistence), resulting in incomplete digestion of lactose and lactose malabsorption in adulthood (1). Secondary forms of lactose malabsorption may be due to inflammation or functional loss of the intestinal mucosa such as celiac disease, infectious enteritis or Crohn's disease. Very rarely, lactase deficiency is congenital due to an autosomal recessive genetic disorder, preventing lactase expression from birth (2). Whereas some people with lactose malabsorption are asymptomatic, most lactose-nonpersisters experience symptoms like abdominal pain, bloating, excess flatulence or diarrhea. Lactose intolerance refers to the syndrome of having one or more symptoms after consumption of lactose-containing food (3). At present, the origin of the symptoms of lactose-intolerance is not well understood.

Several studies have indicated a poor correlation between lactose maldigestion and symptoms of lactose intolerance (4). In a study by Vonk et al. (2003), lactose intolerant subjects with severe symptoms (diarrhea) and intolerant subjects with only mild symptoms (without diarrhea) did not differ in degree of lactose digestion in the small intestine indicating a similar lactase activity and leading them to the hypothesis of a "colon resistence factor" (5). It was suggested that the colonic processing of maldigested lactose may play a role in the symptoms experienced by lactose intolerant patients. When lactose is malabsorbed and enters the colon, it is rapidly fermented by the resident microbiota into a variety of metabolites including lactate, formate, succinate and short chain fatty acids (SCFA, acetate, propionate, butyrate) as well as gases (H2, CO2 and CH4). When incubating fecal samples from lactose-tolerant and intolerant subjects with lactose, the samples from the lactose-intolerant subjects showed faster production rates of D- and L-lactate, acetate, propionate and butyrate, as compared to tolerant subjects (6). Although the colon is thought to possess a high capacity to absorb SCFA, it was hypothesized that a temporary accumulation of these metabolites due to rapid fermentation of maldigested lactose could be responsible for abdominal pain, excess flatulence and bloating (7;8). Possible mechanisms proposed to explain how SCFA might induce symptoms included an increase in the osmotic load that draws fluid to the colonic lumen, changes in colonic motility and an increased colonic sensitivity (9-11). However, the calculated amount of fluid drawn in the colon is unlikely to cause symptoms considering the high water absorbing capacity of the colon and the effect of SCFA on colonic motility and colonic sensitivity have only been observed in rats and not in humans.

More recently, Campbell et al. introduced the bacterial metabolic toxin hypothesis, stating that also other bacterial metabolites, such as alcohols, aldehydes, acids and ketones, resulting from carbohydrate fermentation play a role in the pathogenesis of lactose-intolerance. These metabolites might inhibit bacterial growth and affect eukaryotic cells (12). In our own previous studies in which we related colonic fermentation patterns to parameters of cytotoxicity, we identified compounds like propionic acid, medium chain fatty acids, 1-octanol and heptanal as more prevalent in the most cytotoxic samples (13), supporting the hypothesis of Campbell et al. Therefore, it seems necessary to include not only SCFA, but also other metabolites, in the investigation of the pathogenesis of lactose intolerance.

Differences in fermentation patterns might be associated with differences in the composition and/or activity of the intestinal microbiota. Evidence on the potential role of the colonic microbiota in lactose intolerance is very limited. Total bacterial numbers were not significantly different between 16 intolerant and 11 tolerant lactose maldigesters although a negative correlation between total bacteria and symptom score was found (14). Similarly, the composition of fecal microbiota was not different between 5 intolerant and 7 tolerant subjects (6).

DETAILED DESCRIPTION:
In this study we will compare colonic fermentation and parameters of gut health (fecal water cytotoxicity) between patients who are lactose intolerant, patients who have lactose malabsorption and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy or positive lactose breath test
* > 18 Year
* 18 kg/m²<BMI<27.5 kg/m²
* regular dietary pattern

Exclusion Criteria:

* intake of antibiotics 1 month prior to sample collection
* abdominal chirurgical intervention except appendectomy
* intake of medication 14 days prior to sample collection
* vegetarian
* intake of pre- or probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a positive test (reduced lactose digestion and increased H2-excretion) and complaints will be included in the group of lactose-intolerant patients and patients with a positive result without complaints will be included in the group of lactose-malabsorption patients. Subjects with a normal breath test will be recruited as controls.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
fecal water genotoxicity | 1 day
  Fecal water, prepared by ultracentrifugation of fecal samples, will be incubated with HT-29 cells, a colonic adenocarcinoma cell line. Fecal water genotoxicity will be assessed using the Comet Assay, a sensitive method to detect DNA damage at the level of the individual eukaryotic cell. During the Comet Assay, the cells undergo electrophoresis causing movement of the damaged DNA out of the nucleus. The amount of DNA damage will be determined by measuring the extent the DNA has moved out of the nucleus, using fluorescent microcropy and dedicated software.

SECONDARY OUTCOMES:
fecal water cytotoxicity | 1 day
  Fecal water cytotoxicity will be measured using the WST-1 assay, a colorimetric test based on the conversion of the tetrazolium salt WST-1 by cellular mitochondrial dehydrogenases present in viable cells. The dilution of fecal water at which 50% of the cells survive will be determined. The higher the dilution, the more cytotoxic the sample is.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Professor, Principal Investigator — KU Leuven
Locations (1):
- TARGID, KU Leuven, Leuven, Vlaams-Brabant, Belgium